CLINICAL TRIAL: NCT05665101
Title: EndoVascular Aortic Repair With Sac Embolization for the Prevention of Type II Endoleaks (the EVAR-SE Study)- A Randomized Controlled Multicentre Study in Germany
Brief Title: EndoVascular Aortic Repair With Sac Embolization for the Prevention of Type II Endoleaks (the EVAR-SE Study)
Acronym: EVAR-SE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Christoph Knappich (Other)
Collaborators: Technical University of Munich (Other); St. Josefs-Hospital Wiesbaden GmbH (Other); University Hospital Augsburg (Other); University Hospital Carl Gustav Carus (Other)
Responsible Party: Sponsor-Investigator, Christoph Knappich, Principal Investigator, Technical University of Munich
Organization: Technical University of Munich (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V1.1; 01KG2128 (Other Grant/Funding Number: Bundesministerium für Bildung und Forschung)
Record Dates: First submitted 2022-12-07; First posted 2022-12-27 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Abdominal Aortic Aneurysm; Endoleak
Keywords: Abdominal Aortic Aneurysm; Endoleak; Endovascular aortic aneurysm repair; Coiling; Endoleak Type II
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Endoleak

STUDY DESIGN:
Intervention Model Description: randomized controlled
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EVAR with SE (Experimental): Patients in the EVAR-SE arm will receive EVAR with additional coil embolization of the aneurysm sac.
  Interventions: Procedure: Coil embolization of aneurysm sac
- standard EVAR (No Intervention): Patients in the standard EVAR arm will receive EVAR without additional coil embolization of the aneurysm sac.

INTERVENTIONS:
Procedure: Coil embolization of aneurysm sac — Patients are treated with standard EVAR with additional coiling of the aneurysm sac. The distinct type of coils used is not predefined.
  Arms: EVAR with SE

SUMMARY:
Beyond a certain threshold diameter, Abdominal aortic aneurysms (AAA) are treated by open surgical repair or, more often by endovascular aortic aneurysm repair (EVAR). The latter involves implantation of a stent-graft and thereby exclusion of the AAA from the blood circuit. Small vessels supplying parts of the bowel or the spine are regularly covered. In a quarter of patients, this may result in an inversion of blood flow in the mentioned vessels, leading to persistent blood flow within the AAA, referred to as type II endoleak (T2EL). Occurrence of T2EL is associated with complications like AAA growth or even rupture.

Secondary interventions to treat T2EL often fail and may be highly invasive. Various risk factors for T2EL have been described. This enables prediction whether a patient is at high risk for T2EL after EVAR. Deployment of metal coils in the aneurysm sac as part of the EVAR procedure can reduce the risk for T2EL.The present study aims to assess the efficacy of sac embolization during EVAR to prevent T2EL.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Infrarenal AAA ≥50 mm maximum diameter
* Indication for EVAR within IFU of company
* Presence of one or both high risk criteria on CT-A: ≥5 patent efferent vessels (inferior mesenteric and/or lumbar artery, and/or median sacral artery) or <40% thrombus at largest AAA diameter

Exclusion Criteria:

* Ruptured AAA
* Fenestrated or branched EVAR
* Concomitant iliac artery aneurysm
* Non-ability to adhere to the FU protocol
* Lack of consent
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-01-15 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Type II Endoleak at 12 months after procedure | 12 months
  Evaluation of the T2EL proportion of the intervention group as compared to the control group at 12 months after EVAR treatment as measured by CEUS and/or CT-A

SECONDARY OUTCOMES:
Type II Endoleak during follow up | 2-4 days
  T2EL 2-4 days after EVAR treatment detected by CEUS and/or CT-A
Type II Endoleak during follow up | 30 days
  T2EL 30 days after EVAR treatment detected by CEUS and/or CT-A
Type II Endoleak during follow up | 6 months
  T2EL 6 months after EVAR treatment detected by CEUS and/or CT-A
Re-intervention | 12 months
  Rates of any re-intervention (for endoleaks, occlusions, graft infection, graft migration)
Type I or III Endoleak | 12 months
  Occurrence of any EL Type I or III
AAA morphology | 12 months
  Changes of AAA diameter as measured by CT-A in comparison to initial CT-A scan at V0
AAA morphology | 12 months
  Changes of AAA volume as measured by CT-A in comparison to initial CT-A scan at V0
AAA rupture | 12 months
  Rate of AAA rupture 12 months after EVAR treatment
Mortality | 12 months
  Mortality (aneurysm-related/not aneurysm related) 12 months after EVAR treatment
life quality | 12 months
  Change in quality of life assessed by SF-36 from baseline to 12 months after EVAR treat-ment

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Knappich, PD Dr. med., Principal Investigator — Technical University Munich
Locations (1):
- TUM Klinikum Rechts der Isar, Klinik und Poliklinik für Vaskuläre und Endovaskuläre Chirurgie, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Knappich C, Kirchhoff F, Fritsche MK, Egert-Schwender S, Wendorff H, Kallmayer M, Haller B, Hyhlik-Duerr A, Reeps C, Eckstein HH, Trenner M. Endovascular aortic repair with sac embolization for the prevention of type II endoleaks (the EVAR-SE study): study protocol for a randomized controlled multicentre study in Germany. Trials. 2024 Jan 2;25(1):17. doi: 10.1186/s13063-023-07888-8. PMID 38167068